CLINICAL TRIAL: NCT05844709
Title: Effectiveness of Nursing Care Bundle for the Prevention of Intraventricular Hemorrhage in Preterm Infants
Status: Completed | Type: Observational
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 202107092RIND
Record Dates: First submitted 2023-02-23; First posted 2023-05-06 (Actual); Last update posted 2023-07-25 (Actual); Status verified 2023-02

CONDITIONS: Intraventricular Hemorrhage of Prematurity; Nursing Caries
Keywords: premature infants; bundle care; Intraventricular hemorrhage (IVH)
MeSH Terms: conditions — Premature Birth

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Control group: The infants will be divided into 200 in the control group. Eligible hospitalized preterm infants that met the inclusion criteria from January 2017 to December 2019 were selected for the control group by retrospective cohort.
- Experimental group: The infants will be divided into 30 in the experimental group.
  Interventions: Other: IVH care Bundle

INTERVENTIONS:
Other: IVH care Bundle — The experimental group received bundle nursing care within 3 days after birth in addition to routine nursing care after consent was given and the informed consent form was signed.
  IVH care Bundle: 1. Maintaining midline head position 2. Avoid prone, place in supine or side-lying position 3. Incubator tilted 15-30 degrees 4. Slow withdrawal and flushing for UAC, UVC, and PAL.
  Groups: Experimental group

SUMMARY:
Existing measures to prevent intraventricular hemorrhage in preterm infants include preventing premature delivery, pre-natal administration of corticosteroid, active treatment of chorioamnionitis, and improvement of postnatal resuscitation and transfer process. Many overseas studies show that nursing care can reduce the risk of intraventricular hemorrhage and death, but there is no such study in Taiwan.

Objective: to explore the effect of bundle nursing care on prevention of IVH in premature infants.

DETAILED DESCRIPTION:
A quasi-experimental study design was employed and a total of 230 preterm infants with birth weight less than 1,500 g or gestational age ≤30 weeks will be recruited at the neonatal intensive care unit of National Taiwan University Hospital. The infants will be divided into 200 in the control group and 30 in the experimental group. Enrollment began after approval was granted by the Institutional Review Board. Eligible hospitalized preterm infants that met the inclusion criteria from January 2017 to December 2029 were selected for the control group by retrospective cohort and matched by the gestational age, birth weight and delivery method with the experimental group. The experimental group received bundle nursing care within 3 days after birth in addition to routine nursing care after consent was given and the informed consent form was signed. The study tools include 1. Intervention Tools: small towel or head positioning pillow (Tortle Midliner) and timer; 2. Data collection: Self-created questionnaire on awareness and behavior for preventing intraventricular hemorrhage in preterm infants in nurses, medical record and bundle care implementation record. The data were analyzed by descriptive statistics, t-test, Chi-square test and Logistic regression using SPSS 26 statistical software. The expected results are reduction in the incidence of intraventricular hemorrhage, the length of stay in the intensive care unit and mortality.

ELIGIBILITY:
Inclusion Criteria:

* Inborn Preterm infants
* Preterm infants with birth weight less than 1,500 g or gestational age ≤30 weeks

Exclusion Criteria:

* Preterm infants with congenital malformations
* Genetic syndromes
* Congenital infections of the TORCHS group(syphilis, rubella, herpes, toxoplasmosis, and cytomegalovirus)
* Resuscitation and Pneumothorax at birth.

Ages: 1 Day to 1 Month | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Very Low Birth Weight(VLBW) : Preterm infants with birth weight less than 1500g.
  Intraventricular hemorrhage (IVH) is one of the serious complications in preterm infants and is present in about 25-30% of VLBW, which is related to long-term neurological sequelae and mortality.
Sampling Method: Probability Sample
Enrollment: 178 (Actual)
Dates: Start 2022-09-10 (Actual); Primary Completion 2023-04-15 (Actual); Study Completion 2023-07-04 (Actual)

PRIMARY OUTCOMES:
The incidence of intraventricular hemorrhage | 72 postnatal hours
  Grading of Intraventricular Hemorrhage
The incidence of intraventricular hemorrhage | 168 postnatal hours
  Grading of Intraventricular Hemorrhage

SECONDARY OUTCOMES:
The length of stay in the intensive care unit | From date of admission until the date of leave Neonatal intensive care unit up to 48 weeks
  Inpatient days
Mortality | From date of admission until the date of death from any cause up to 4 postnatal weeks
  neonatal death

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Fu-Chang Tsai, Study Chair — National Taiwan University Hospital
Locations (1):
- Peiyi ,Lu, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No